CLINICAL TRIAL: NCT02782234
Title: Application of Contract Management Mode in Maintaining Body Fluid Balance of Peritoneal Dialysis Patients
Brief Title: Application Contract Management Mode in Maintaining PD Fluid Balance
Acronym: ACMMPDFB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Li Liu, Supervisor nurse, The Second Affiliated Hospital of Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2 ndharbinmu
Record Dates: First submitted 2016-04-08; First posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Contract Management PD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- not contract management (No Intervention): monthly follow-up phone or family visit completed as regulation, and instruct them proper healthy training.
- Contract management (Experimental): In accordance with the contract content, researchers and participants should manage and maintain the liquid balance of the participants. Signed doctors and nurses should undergo the follow-up phone or family visit on time, instruct them proper healthy training, and provided necessary information data. By telephone, SMS, wechat, remind and urge the participants to take the lifestyle and behavior regulate in the contract. Participants should supervise and manage the fluid unbalance (Edema, hypertension, heart failure, and fluid imbalance of intake and output etc.), and feedback the Management and supervision to researchers according to contract.
  Interventions: Behavioral: Contract management

INTERVENTIONS:
Behavioral: Contract management
  Arms: Contract management

SUMMARY:
Contract management is a new management mode.

To help patients achieve fluid balance through contract management, that is:

1. edema, congestive heart failure and other similar symptoms begin to reduce to disappear;
2. Blood pressure control in normal range, that is 90-140/60-90mmHg, or the target value prescribed by the doctors；
3. Fluid intake and output keep in balance;
4. No imbalance symptoms turn out, such as edema, congestive heart failure, etc.

DETAILED DESCRIPTION:
Contract management is a new management mode, it stipulate and constraint various relationship by various duties, institutions and regulations.

To help patients achieve fluid balance through contract management, that is:

1. edema, congestive heart failure and other similar symptoms begin to reduce to disappear;
2. Blood pressure control in normal range, that is 90-140/60-90mmHg, or the target value prescribed by the doctors；
3. Fluid intake and output keep in balance;
4. No imbalance symptoms turn out, such as edema, congestive heart failure, etc.

In addition to help keeping the fluid balance through contract balance, but also:

1. Improve compliance;
2. Improve the patients' cognition of fluid balance;
3. Improve the ability of self-management of fluid balance.

ELIGIBILITY:
Inclusion Criteria:

1. Older or equal to 18 years, younger or equal to 65 years, CAPD duration over 6 months
2. Edema or congestive heart failure happen
3. Patients with poor control of blood pressure, that is less than 90/60mmHg,or over 140/90mmHg, or the Bp does not meet the value given by doctors
4. Patients with fluid imbalance of intake and output.

Exclusion Criteria:

1. Younger than 18, or older than 65, or CAPD period less than 6 months
2. The primary disease is high blood pressure, or edema due to low protein
3. Patients that lost control of daily life
4. Malignant tumor or pregnancy
5. Falling in Chronic infection or severe complication within 1 month, such as hepatic disease, hemorrhage of digestive tract, etc.
6. Patients with cognition impairment, conscious disorder, or mental disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Volume of fluid intake and output keep in balance measured in ml. | 24 hours
  as the physiological parameter for this Outcome. Volume measurement unit should be used in pd subjects, the unit ml.
Change in Blood Pressure | two times a day, through study completion, an average of 6 months. changed from baseline
  two times a day, blood pressure measure at a.m.6∶0 0～ 8∶0 0 ,p.m.15∶0 0～ 18∶0 0. The subjects for the first time measuring blood pressure for the baseline.
Change in weight | once a day, through study completion, an average of 6 months. changed from baseline
  The subjects for the first time measuring weight for the baseline measured in kg.

IPD SHARING:
Plan to Share IPD: No